CLINICAL TRIAL: NCT00939536
Title: Studies in Fasted Healthy, Normal Subjects to Compare the Single Dose Bio-availability of Torrent's Zolpidem Tartrate Tablets 10 mg and Sanofi-Synthelabo's Ambien® 10 mg Tablets
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Ltd.'s Zolpidem Tartrate Tablets Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: US/05/003
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Torrent's Zolpidem Tartrate Tablets 10 mg (Experimental): Normal Healthy Human Subjects receiving Torrent's Zolpidem Tartrate Tablets 10 mg
  Interventions: Drug: Zolpidem Tartrate Tablets 10 mg
- Sanofi-Synthelabo's Ambien® 10 mg Tablets (Active Comparator): Normal Healthy Human Subjects receiving Sanofi-Synthelabo's Ambien® 10 mg Tablets
  Interventions: Drug: Zolpidem Tartrate Tablets 10 mg

INTERVENTIONS:
Drug: Zolpidem Tartrate Tablets 10 mg

SUMMARY:
* Objective:

  * To compare the rate and extent of absorption of Zolpidem Tablets 10mg: Test Product: Zolpidem Tablets 10mg manufactured by Torrent Pharmaceuticals Limited, India Reference Product: Ambien® Tablets 10 mg (Reference Listed Drug) manufactured by Sanofi- Synthelabo Inc. under fasting conditions in 24 healthy, adult, human subjects.
* Study Design:

  * Open label, randomized, two-period, two-treatment, two-sequence single dose crossover design.

DETAILED DESCRIPTION:
Open label, randomized, two-period, two-treatment, two-sequence single dose

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects in the range of 18 - 45 years of age.
2. Body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart. (Appendix A)
3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and body temperature)
4. Subjects with normal findings as determined by hematological tests, serum chemistry, urine analysis, ECG and X-ray.
5. Willingness to follow the protocol requirement as evidenced by written, informed consent.
6. Agreeing to, not using any medication (prescription and over the counter), including vitamins and minerals for 15 days prior to study and during the course of the study.
7. No history or presence of significant alcoholism or drug abuse in the past one year.
8. Non-smokers, ex smokers and light smokers will be included. "Light smokers are defined as someone smoking 10 cigarettes or less per day, ex smokers as someone who completely stopped smoking for at least 3 months.

Exclusion Criteria:

1. Requiring medication for any ailment including enzyme-modifying drugs Use of any drugs known to induce or inhibit hepatic drug metabolism (e.g.s, inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors: SSRIs, cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
2. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
3. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic diseases.
4. History of psychiatric disorder or history of suicide attempt.
5. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
6. History of malignancy or other serious diseases.
7. Refusal to abstain from food for ten (10) hours prior to study drug administration the day of each study period and for four (4) additional hours each, post dose.
8. Refusal to abstain from water for one (1) hour prior to study drug administration the day of each study period and for two (2) additional hour, post dosing.
9. Any contraindication to blood sampling.
10. Refusal to abstain from smoking or consumption of tobacco products 24 hours before dosing until last sample collection of each period. Habituation of tobacco necessitating uninterrupted tobacco consumption.
11. Use of xanthine-containing beverages or food for 48 hours prior to each drug dose.
12. Blood donation 90 days prior to the commencement of the study.
13. Subjects with positive HIV tests, HbsAg or Hepatitis-C tests.
14. Known history of allergic reactions to zolpidem or other related drugs.
15. History of drug abuse in the past one year.
16. Use of prescription medication within 14 days prior to administration of study medication or over the counter products (including natural food supplements, vitamins, garlic as a supplement) within 2 weeks prior to administration of study medication, except for topical products without systemic absorption.
17. Pregnant and lactating women.

    * At the time of screening, prior to enrollment, presence of pregnancy will be confirmed by urine pregnancy test.
    * Female subjects not confirming to using birth control measures, from the date of screening till the completion of the second period of the study. Abstinence, barrier methods (condom, diaphragm, etc.) are acceptable. Use of hormonal contraceptives either oral or implants will not be acceptable.
18. Female subjects whose menstruation cycle coincides with the study periods.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Accutest Research Laboratories Pvt. Ltd., Mumbai, Maharashtra, India

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: healthy, normal subjects
Groups:
- Torrent's Zolpidem First, Then Ambien: For period one - on the morning of Day 1 subjects received Torrent's Zolpidem 10 mg.
  Followed by a 7 day washout period.
  For period two - on the morning of Day 1 subjects received the reference formulation, Ambien 10 mg.
- Ambien First, Then Torrent's Zolpidem: For period one - on the morning of Day 1 subjects received the reference formulation, Ambien 10 mg
  Followed by a 7 day washout period.
  For period two - on the morning of Day 1 subjects received the test formulation, Torrent's Zolpidem 10 mg.
Period: First Intervention
Arm/Group | Torrent's Zolpidem First, Then Ambien | Ambien First, Then Torrent's Zolpidem
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Torrent's Zolpidem First, Then Ambien | Ambien First, Then Torrent's Zolpidem
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Torrent's Zolpidem Tartrate Tablets 10 mg
- Active Comparator: Ambien® 10mg tablets
- Total: Total of all reporting groups
Arm/Group | Experimental | Active Comparator | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.7) | 28.2 (6.7) | 28.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  India | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma
Time Frame: plasma samples were obtained from blood drawn at 0 (within 60 minutes prior to dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 20 and 24 hours (18 samples) after administration of the dose.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 24 | 24
ng/ml | 177.69 (57.05) | 172.64 (72.15)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 24 | 24
mcg*hr/mL | 751.31 (399.17) | 717.71 (401.92)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity AUC(0-∞)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Experimental | Active Comparator
Number analyzed (Participants) | 24 | 24
mcg*hr/mL | 778.16 (418.74) | 741.65 (415.73)

ADVERSE EVENTS:
Arm/Group | Experimental | Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 9/24 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Experimental (N=24) | Active Comparator (N=24)
vomiting (General disorders) | 4 (4) | 0/0 (0)
nausea (General disorders) | 2 (2) | 0/0 (0)
regurgitation of water content (General disorders) | 2 (2) | 0/0 (0)
giddiness (General disorders) | 1 (1) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other